CLINICAL TRIAL: NCT02223819
Title: Phase II Trial of Adjuvant Crizotinib in High-Risk Uveal Melanoma Following Definitive Therapy
Brief Title: Crizotinib in High-Risk Uveal Melanoma Following Definitive Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAO8010
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Uveal Melanoma
Keywords: Crizotinib; 14-063
MeSH Terms: conditions — Uveal Melanoma | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Crizotinib (Experimental): Subjects will receive 48 weeks (12 four-week cycles) of crizotinib 250 mg PO twice a day (BID). Subjects will be evaluated by routine bloodwork and physical exam every 4 weeks while they are receiving crizotinib and during follow up period.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — An anti-cancer drug acting as an anaplastic lymphoma kinase (ALK) and c-ros oncogene 1 (ROS1) inhibitor, used to treat non-small cell lung cancer (NSCLC) that has spread to other parts of the body and is caused by a defect in a gene called ALK.
  Crizotinib will be provided as capsules containing 200 or 250 mg of study medication for oral administration.
  Other Names: Xalkori

SUMMARY:
The study is designed to determine the 32 month rate of distant relapse in patients with uveal melanoma who are at high risk of recurrence following definitive therapy with surgery or radiation who receive adjuvant crizotinib; and secondarily, the overall survival and disease specific survival in this patient population.

DETAILED DESCRIPTION:
Uveal melanoma is the most common primary intraocular malignancy in adults, and arises from melanocytes within the choroid plexus of the eye. Melanomas of the ocular and adnexal structures comprise approximately 5% of all melanomas and are biologically and prognostically distinct from cutaneous melanoma. In the United States, an estimated 2000 patients are diagnosed with this disease each year.

The development of metastasis in this disease is common and occurs in approximately 50% of patients with posterior uveal melanoma within 15 years after the initial diagnosis and treatment. Uveal melanoma is thought to be particularly resistant to systemic treatment, and no systemic therapy has yet been demonstrated to improve survival. Drugs commonly used to treat advanced cutaneous melanoma rarely achieve durable responses in patients with uveal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of uveal melanoma at least 12 mm in largest basal diameter as clinically determined by the treating investigator. Cytologic determination of diagnosis is not required. Size is based on clinical assessment (e.g. by ultrasound or direct ophthalmoscopy) prior to enucleation or radiation therapy.
* Definitive therapy of the primary uveal melanoma must have been performed within 90 days of initiating protocol therapy.
* High-risk (class 2) uveal melanoma as determined by gene expression profiling
* No evidence of metastatic disease.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (Karnofsky ≥ 70%.
* Life expectancy of greater than 3 months.
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count (ANC) >1,000 cells/mm³
* Platelet count >75,000/mm³
* Hemoglobin >9.0g/dL
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) <3x upper limited of normal (ULN)
* Total bilirubin <2x ULN
* Alkaline phosphatase <3x ULN
* Serum creatinine <2x ULN or a creatinine clearance > 60mL/min
* Note: Patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert syndrome) will be eligible at the discretion of the treating physician and/or the principal investigator.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation until 4 months after completion of crizotinib administration. Women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study therapy, and 4 months after completion of crizotinib administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of another malignancy except for those who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies not requiring active therapy, are eligible. Consult the study Principal Investigator if unsure whether second malignancies meet the requirements specified above.
* Any major surgery or extensive radiotherapy (except that which is required for definitive treatment of primary uveal melanoma), chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to initiation of study therapy.
* History of prior crizotinib use.
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study therapy and during the study.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to crizotinib.
* Concurrent administration of crizotinib and a strong inhibitor or inducer of CYP3A is not permitted. Many over-the-counter and dietary supplements also inhibit or induce CYP3A and thus are prohibited.
* A QT interval corrected for heart rate using the Bazett's formula QTcB ≥ 480 msec.
* Concurrent administration of crizotinib and agents that can cause QTc prolongation is not permitted.
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection, which will be allowed). HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with crizotinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaheer A Khan, DO, Principal Investigator — Assistant Professor of Medicine at the Columbia University Medical Center
Locations (4):
- United States (4):
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Columbia Univeristy Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib: Subjects will receive 48 weeks (12 four-week cycles) of crizotinib 250 mg PO twice a day (BID). Subjects will be evaluated by routine bloodwork and physical exam every 4 weeks while they are receiving crizotinib and during follow up period.
  Crizotinib: An anti-cancer drug acting as an anaplastic lymphoma kinase (ALK) and c-ros oncogene 1 (ROS1) inhibitor, used to treat non-small cell lung cancer (NSCLC) that has spread to other parts of the body and is caused by a defect in a gene called ALK.
  Crizotinib will be provided as capsules containing 200 or 250 mg of study medication for oral administration.
Period: Overall Study
Arm/Group | Crizotinib
Started | 34
Completed | 32
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Crizotinib
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 60 [26 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25
  Hispanic | 2
  Other/Unknown | 7
Region of Enrollment [Number; unit: participants]
  United States | 34
Largest basal diameter [Median (Full Range); unit: mm] — A larger basal diameter generally indicates more advanced disease.
  mm | 14.0 [12 to 21]
Eastern Cooperative Oncology Group (ECOG) Status [Median (Full Range); unit: units on a scale] — ECOG is a performance status scale used to assess functional status. The scale ranges from 0 (Fully active) to 5 (Dead) with a higher score indicating a worse outcome.
  units on a scale | 0 [0 to 1]

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival (RFS) Rate at 32 Months
Description: RFS rate will be defined as the percentage of patients who do not experience any new tumor growth at any site on the body distant from the primary site or death from any cause from the time of study entry to the end of the relevant timepoint. RFS probabilities were estimated using Kaplan-Meier method.
Time Frame: 32 Months
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Crizotinib
Number analyzed (Participants) | 32
Probability | 50 [33 to 67]

2. Secondary Outcome: Overall Survival (OS)
Description: OS will be defined as the time from treatment start to date of death or last followup. Participants were followed up to 36 months after treatment start and Kaplan-Meier survival analysis was used to generate the Overall Survival estimate.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib
Number analyzed (Participants) | 32
months | 68.3 [51.0 to NA] — The upper limit is not applicable due to limited overall survival events at later timepoints.

3. Secondary Outcome: Disease-Specific Survival (DSS) Time
Description: DSS is defined as the time from treatment start to death due to disease or last followup. Participants who die from other causes will be censored.
Time Frame: Up to 36 months
Population: Data needed for for DSS calculation (death due to disease) was not collected as participants were no longer actively followed at the time of death.
Arm/Group | Crizotinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Treatment Discontinuation Due to Toxicity
Description: Toxicity grading will be performed in accordance with NCI CTCAE, version 4.0.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib
Number analyzed (Participants) | 32
Participants | 4

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Crizotinib
All-Cause Mortality (participants affected / at risk) | 11/34
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crizotinib (N=34)
Myocardial infarction (Cardiac disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Left leg and upper back squamous cell carcinomas in situ (Skin and subcutaneous tissue disorders) | 1 (1)
Overdose (General disorders) | 1 (1)
Potential new cancer left renal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crizotinib (N=34)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 13 (31)
Alkaline phosphatase increased (Investigations) | 6 (8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (14)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 16 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Elevated liver enzymes (Blood and lymphatic system disorders) | 2 (3)
Blurred vision (Eye disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (4)
Constipation (Gastrointestinal disorders) | 12 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Creatine phosphokinase (CPK) Increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 8 (18)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 21 (48)
Dizziness (Nervous system disorders) | 11 (13)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 6 (6)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (9)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Edema limbs (General disorders) | 12 (13)
Edema trunk (General disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Fatigue (General disorders) | 18 (30)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Flashing lights (Eye disorders) | 4 (6)
Flatulence (Gastrointestinal disorders) | 2 (2)
Floaters (Eye disorders) | 6 (6)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait disturbance (General disorders) | 1 (4)
Gastritis (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Glaucoma (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1)
Elevated Lactate Dehydrogenase (LDH) (Hepatobiliary disorders) | 12 (14)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (30)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (10)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (12)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (30)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (18)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
Hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Localized edema (General disorders) | 5 (6)
Lymphedema (Vascular disorders) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (4)
Malaise (General disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 19 (24)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (3)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (4)
Presyncope (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (5)
Renal calculi (Renal and urinary disorders) | 1 (1)
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scleral disorder (Eye disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 15 (21)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (2)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Uterine infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 7 (7)
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 1 (1)
Cataract surgery (Investigations) | 1 (1)
Colonoscopy (Investigations) | 1 (1)
Elevated transaminases (Hepatobiliary disorders) | 1 (1)
Endoscopy (Investigations) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2)
Herpes Zoster (Skin and subcutaneous tissue disorders) | 1 (1)
Hypochloremia (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoproteinemia (Investigations) | 2 (2)
Intermittent visual disturbance, left eye (Eye disorders) | 1 (1)
Interstitial lung disease (Investigations) | 1 (1)
Kidney pain with pressure during urination (Renal and urinary disorders) | 1 (1)
Left Hip Pain (Investigations) | 1 (1)
Leukopenia (Investigations) | 1 (1)
Migraine (Nervous system disorders) | 1 (2)
Neutrophil count increased (neutrophilia) (Investigations) | 1 (1)
Palinopsia (Eye disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary embolus (Vascular disorders) | 1 (1)
Shortness of breath (Investigations) | 1 (1)
Uncontrolled Diarrhea (Gastrointestinal disorders) | 1 (1)
Vision loss (Eye disorders) | 1 (1)
Visual disturbances (Eye disorders) | 1 (1)
Visual disturbances (double vision) (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT02223819/Prot_SAP_000.pdf